CLINICAL TRIAL: NCT06580951
Title: Regenerative Peripheral Nerve Interface for Prophylaxis Against Post-Breast Surgery Pain
Brief Title: Regenerative Peripheral Nerve Interface for Prophylaxis Against Post-Breast Surgery Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Kokosis (Other)
Responsible Party: Sponsor-Investigator, George Kokosis, Associate Professor, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24042301
Record Dates: First submitted 2024-08-08; First posted 2024-08-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Post-mastectomy Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Masking Description: Those who agree and sign the informed consent form will be randomized in 1:1 fashion (50/50 chance) to either the RPNI group or the no RPNI (Control) group. Subjects will remain blinded to their assigned study arm until their study participation has concluded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPNI (Experimental): Subjects will complete BREAST-Q Pre-Op (Qol) survey and Pain Distribution survey prior to Surgery. Subjects will in the RPNI arm will undergo mastectomy with breast reconstruction surgery with regenerative peripheral nerve interface. Subjects will complete BREAST-Q Post-Op (QoL) survey and Pain Distribution Survey at Months 1, 3, 6, and 12 post-surgery. Information about the patient and course of care will be collected from electronic medical records.
  Interventions: Procedure: Regenerative Peripheral Nerve Interface
- No RPNI (Control) (No Intervention): Subjects will complete BREAST-Q Pre-Op (Qol) survey and Pain Distribution survey prior to Surgery. Subjects undergo mastectomy with breast reconstruction surgery without regenerative peripheral nerve interface. Subjects will complete BREAST-Q Post-Op (QoL) survey and Pain Distribution Survey at Months 1, 3, 6, and 12 post-surgery. Information about the patient and course of care will be collected from electronic medical records.

INTERVENTIONS:
Procedure: Regenerative Peripheral Nerve Interface — The RPNI portion of the case will consist of blunt dissection of the cut sensory branches of the intercostal nerves at the T3 and/or T4 levels, with creation of a peripheral nerve interface using a small cuff of dissected pectoralis muscle and 3-0 Monocryl suture. The breast reconstruction will otherwise be performed as per standard protocol.
  Arms: RPNI

SUMMARY:
Regenerative peripheral nerve interface (RPNI) was first developed in 2012 by Dr. Paul Cederna at the University of Michigan as a means for amputees to control their prothesis with their minds. In the decade that followed, it was found RPNI surgery not only provided amputees with neuroma (a growth made up nerve tissue) pain relief but could help prevent neuroma from developing as well.

This single center, randomized controlled, investigator-initiated study will look at whether the RPNI, a nerve burying procedure involving protecting sensory nerves with a small piece of the patient's pectoralis muscle, performed at the time of the standard mastectomy with immediate breast reconstruction surgery can prevent and/or reduce the risk for long-term nerve pain after breast cancer surgery (also called neuroma-related post-breast surgery pain syndrome (PBSPS)) versus the standard surgery alone (Control group). Symptoms of PBSPS include discomfort, numbness, tingling, and shooting pain in the chest and breast area. It is relatively common and may have many causes.

About 200 adult females (18-65 years old) who are scheduled to undergo mastectomy with immediate breast reconstruction surgery will be approached for this study. Those who agree and sign the informed consent form will be randomized in 1:1 fashion (50/50 chance) to either the RPNI group or the no RPNI (Control) group. Study participants will complete self-reported surveys (pre-surgery and at Months 1, 3, 6, and 12 post-surgery) designed to measure pain levels, quality of life, and function before and after surgery. Study participation will last approximately 12 months. Subjects will remain blinded to their assigned study arm until their study participation has concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female 18 to 65 years of age.
2. Undergoing breast mastectomy with immediate reconstruction.
3. Able to provide informed consent and comply with study procedures.

Exclusion Criteria:

1. History of chronic pain syndrome unrelated to breast surgery.
2. Unwillingness or inability to comply with the study's follow-up requirements.
3. Cognitive impairment or language barriers preventing proper understanding of study procedures and assessments.
4. Participation in other interventional trials or treatments aimed at pain management that could confound study outcomes as determined by the PI.
5. Other medical or surgical contraindication to the involved procedure (RPNI) as determined by the PI.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Recruitment is limited to females as virtually all cases of breast cancer, and associated mastectomy and reconstruction procedures, are in women.
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of neuroma-related PBSPS | 12 months
  The study's primary endpoint will be the incidence of neuroma-related PBSPS, assessed by comparing the proportion of participants in each group who experience this condition during a follow-up period of 12 months, through review of electronic medical records.

SECONDARY OUTCOMES:
Quality of Life change | 12 months
  This endpoint will be evaluated through use of the Breast-Q questionnaires.The Breast-Q questionnaire is a type of standardized patient-reported outcomes form. There is no overall or total BREAST-Q score, only scores for each independent scale. All BREAST-Q scales are transformed into scores that range from 0-100. The scores are computed by adding the response items together and then converting the raw sum scale score to a score from 0-100. For all BREAST-Q scales, a higher score means greater satisfaction or better QOL (depending on the scale). If missing data is less than 50% of the scale's items, study team will use the mean of the completed items. Study team will convert the raw summed scale score into a score from 0 (worst) to 100 (best).
Safety and Adverse Events | 12 months
  The electronic medical record will be reviewed and any safety or adverse events adjudicated and recorded.
Pain change | 12 months
  Pain Distribution is a peer-reviewed survey that provides a visual reference of various pain distributions of common pathologies affecting the breast, chest, back, and upper extremities, including neuroma-related breast pain, which will allow delineation of the specific etiology causing the patient's pain. For each of the regions surveyed (Underneath Breast, Axilla/Armpit, Radiatin from Chest to Arm, Upper Outer Shoulder, Anterior Shoulder and Axilla/Armpit, Posterior Neck and Shoulder, Posterior Neck Radiating to Arm, Shoulder Blade/Scapula) subjects indicate pain severity and frequency. There is no overall score for the entire survey. The pain severity scale ranges from 0-10. Zero (0) indicates no pain (best), and 10 (ten) indicates the worst pain imaginable (worst). The pain frequency scale ranges from <1 day/week (best) to 7 days/week (worst).

CONTACTS AND LOCATIONS:
Overall Officials: George Kokosis, MD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No